CLINICAL TRIAL: NCT07230080
Title: Efficacy and Safety of Sequential TACE-SBRT Combined With Targeted Immunotherapy in Patients With Intermediate to Advanced Hepatocellular Carcinoma
Brief Title: Sequential TACE-SBRT Combined With Targeted Immunotherapy for Patients With Intermediate to Advanced Liver Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-159
Record Dates: First submitted 2025-09-27; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HCC - Hepatocellular Carcinoma; SBRT; TACE; Immunotherapy; Targeted Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sequential TACE-SBRT With Targeted Immunotherapy Group

SUMMARY:
The goal of this clinical trial is to evaluate whether sequential transarterial chemoembolization (TACE) followed by stereotactic body radiotherapy (SBRT) combined with targeted immunotherapy is effective and safe for patients with intermediate to advanced hepatocellular carcinoma (HCC) who are not eligible for curative treatment such as surgery or liver transplantation.

This is a single-center, single-arm, retrospective study. All participants included in the analysis will have received the combined treatment regimen.

The main question the study aims to answer is:

Can sequential TACE-SBRT combined with targeted immunotherapy improve the objective response rate (ORR) in patients with intermediate to advanced HCC?

Interventions

Participants in this study have undergone the following treatments:

TACE: a minimally invasive procedure to block the blood supply to the tumor while delivering chemotherapy directly.

SBRT: a highly precise form of radiation therapy targeting the liver tumor. Targeted immunotherapy: systemic treatment that stimulates the immune system to recognize and attack cancer cells.

Participant Population The study includes adult patients diagnosed with intermediate to advanced HCC who were not candidates for curative resection or transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Unresectable hepatocellular carcinoma (HCC)
* CNLC stage IIb-IIIb
* Target lesion(s) not previously treated with local therapy
* Child-Pugh class A5-B7 liver function
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2
* At least one measurable lesion based on modified RECIST (mRECIST) criteria

Exclusion Criteria:

* Diagnosis of any malignant disease other than primary liver cancer within 3 years prior to enrollment
* Currently participating in another interventional clinical study
* History of allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
* Presence of any severe or uncontrolled systemic disease
* Any medical history, comorbid condition, treatment, or abnormal laboratory finding that may interfere with study results or hinder full participation, or any other situation that the investigator considers inappropriate for enrollment
* Investigator's judgment of other potential risks making the patient unsuitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate to advanced hepatocellular carcinoma (HCC) who received sequential TACE-SBRT followed by targeted immunotherapy at a single tertiary medical center. Eligible participants were adults (≥18 years) with unresectable disease not suitable for curative surgery or liver transplantation, with preserved liver function and measurable lesions. The population represents a hospital-based cohort identified from medical records rather than a community sample.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) according to mRECIST | At baseline and every 3 months after treatment initiation, up to study completion (an average of 6months)
  Objective response rate (complete response + partial response) assessed by mRECIST based on imaging evaluation.

SECONDARY OUTCOMES:
Overall Survival (OS) | From treatment initiation until death from any cause, up to study completion (an average of 26 months)
Progression-Free Survival (PFS) according to mRECIST | From treatment initiation until disease progression or death, whichever occurs first, up to study completion (an average of 15 months)
  Time from treatment initiation to disease progression or death, assessed by mRECIST.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From treatment initiation through study completion, up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hosptial, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No